CLINICAL TRIAL: NCT06645873
Title: Comparison of Continuous Glucose Monitoring and Point-of-Care Measurements on the Intensive Care Unit: An Exploratory Study
Brief Title: Exploration of Continuous Glucose Monitoring on the Intensive Care Unit
Acronym: CGM-IC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kim Kamphorst (Other)
Collaborators: DexCom, Inc. (Industry); Pioneers in Healthcare (Unknown)
Responsible Party: Sponsor-Investigator, Kim Kamphorst, Principal Investigator, Deventer Ziekenhuis
Organization: Deventer Ziekenhuis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL87243.100.24
Record Dates: First submitted 2024-10-03; First posted 2024-10-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-02

CONDITIONS: Hypoglycemia, Hyperglycemia
Keywords: Intensive care units; insulin; Continuous Glucose Monitoring
MeSH Terms: conditions — Hypoglycemia; Hyperglycemia; Insulin Resistance | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Continuous glucose monitoring (Experimental)
  Interventions: Device: Continuous glucose monitoring (CGM) device

INTERVENTIONS:
Device: Continuous glucose monitoring (CGM) device — All included study participants recieve a CGM sensor (Dexcom G7) to monitor blood glucose. The treatment team is blind for the CGM values; the gold standard for glucose control (POC interval measures) will be followed.

SUMMARY:
Both hyperglycemia and hypoglycemia in patients at the intensive care unit (ICU) are strongly associated with increased morbidity and mortality. Accurate and timely measurements of glucose levels in this population are therefore crucial. Continuous glucose monitoring (CGM) appears promising for this purpose, but it is not yet used in the ICU due to insufficient knowledge about its reliability in critically ill patients. The aim of this study is to investigate the discrepancy between CGM and point-of-care measurements in ICU patients and whether this discrepancy is consistent across all ICU patient groups/characteristics.

This study investigates whether continuous glucose monitoring can be used in the intensive care setting.

DETAILED DESCRIPTION:
Hyperglycemia is present in up to 50% of patients admitted to an intensive care unit (ICU) and is strongly associated with elevated morbidity and mortality rates. Therefore, it is important to monitor glucose levels closely. In the ICU, glucose monitoring primarily relies on periodic measurements through point-of-care (POC) meters, which involve invasive blood sampling from venous or arterial lines. To maintain blood glucose concentrations within acceptable ranges, a possible improvement is continuous glucose monitoring (CGM), which is now used to manage glucose levels in diabetic patients in general settings and has shown significant benefits. Studies on the use of CGM in the ICU setting are limited. If CGM reliably measures glucose levels in critically ill patients, it enables earlier intervention and might help to predict hypo- or hyperglycemia based on measurement trends.

Objective: To investigate the discrepancy between CGM and POC measurements in insulin-dependent ICU patients and to study whether these potential discrepancies between CGM and POC vary across patient-related factors, like gender, age, comorbidities, medication use, disease severity scores, treatment in ICU.

Study design: Prospective, multi-centre, single-arm intervention, exploratory study

Intervention: All study participants receive one CGM sensor to monitor glucose levels. A second CGM sensor will only be applied if the first CGM sensor needed to be replaced within 8 days after insertion. The measurements will be blinded to all except the research team.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU
* Insulin-dependent as defined in local protocol
* Age: ≥ 18 y
* Expected length of stay in ICU more than 2 days

Exclusion Criteria:

* Pregnancy
* No informed consent
* Therapeutic hypothermia (less than 34 degrees celsius)
* Platelet count less than 50,000/μL at time of inclusion
* Use of hydroxyurea
* Use of acetaminophen more than 4 g/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Discrepancy glucose CGM - POC | From enrollment until the completion of the continuous glucose monitoring (CGM) placement at 10 days.
  Discrepancy between glucose levels (in mmol/L) measured with Continuous Glucose Monitoring (measured with the Dexcom G7 sensor) and Point-Of-Care (measured with the Accu-check) measurement in insulin-dependent Intensive Care Unit patients.
  The discrepancy is defined as the difference in absolute glucose levels in arterial blood samples.
Variation discrepancy across patient-related factors | From enrollment until the completion of the continuous glucose monitoring (CGM) placement at 10 days.
  The variation of the potential difference in glucose levels (in mmol/L) between CGM (measured with the Dexcom G7 sensor) and POC (measured with the Accu-check) will be analyzed among the following patient-related factors:
  Age at the time of inclusion (in years). Body Mass Index (BMI) (in kg/m²). Gender (Male/Female).
  Comorbidities:
  Hypertension (Yes/No). Hypotension (Yes/No). Pre-existing diabetes (Yes/No). Edema (measured as weight gain in kg). Acidosis (pH value, continuous scale).
  Medication use:
  Corticosteroids (Yes/No). Inotropics (Yes/No and dosage in µg/kg/min). Vasopressors (Yes/No and dosage in µg/kg/min). APACHE II score (Scale). SOFA score (Scale). Reason for ICU admission (Categorical variable, e.g., sepsis, trauma, etc.). Length of ICU stay (in days). Duration of mechanical ventilation (in hours or days). Dialysis (Yes/No).

SECONDARY OUTCOMES:
Adverse events | From enrollment until the completion of the continuous glucose monitoring (CGM) placement at 10 days.
  The number of reported adverse events, such as infections, bleeding, and decubitus, linked to the continuous glucose sensor (Dexcom G7)
Number of missed hypo- and hypreglycemia episodes | From enrollment until the completion of the continuous glucose monitoring (CGM) placement at 10 days.
  The number and percentage of missed hypoglycemia episodes (defined as a glucose level < 4.0 mmol/L) and hyperglycemia episodes (defined as a glucose level > 10 mmol/L), as indicated by the continuous glucose monitoring (CGM) using the Dexcom G7 sensor, were not detected by point-of-care (POC) interval measurements with the Accu-Chek device.
Delay in detection hypo- or hyperglycemia episodes | From enrollment until the completion of the continuous glucose monitoring (CGM) placement at 10 days.
  The time in minutes between the onset of hypoglycemia (defined as a glucose level < 4.0 mmol/L) or hyperglycemia (defined as a glucose level > 10 mmol/L) detected by the continuous glucose monitoring (CGM) using the Dexcom G7 sensor and its subsequent detection via point-of-care (POC) testing with the Accu-Chek device.
Insertion CGM: time till reliable data and lasting time | From enrollment until the completion of the continuous glucose monitoring (CGM) placement at 10 days.
  The duration of time, in minutes, it takes for the CGM (Dexcom G7 sensor) to reliably measure the glucose (defined as MARD <14%) after the sensor is inserted. Duration of time, in hours, the CGM reliably measures the glucose (defined as MARD <14%) after the sensor is inserted.
Impact radiologic procedure | From enrollment until the completion of the continuous glucose monitoring (CGM) placement at 10 days, but only if a radiologic procedure is performed
  The difference in discrepancies between glucose levels (in mmol/L) measured by continuous glucose monitoring (CGM) using the Dexcom G7 sensor and point-of-care (POC) testing with the Accu-Chek device following radiologic procedures (e.g., CT scans and X-rays) is evaluated.
  Discrepancy is defined as the difference in absolute glucose levels in arterial blood samples measured with the POC compared to the continuous glucose levels measured with the CGM.
Location GCM sensor | From enrollment until the completion of the continuous glucose monitoring (CGM) placement at 10 days.
  The difference in mean absolute relative difference (MARD) between glucose levels (in mmol/L) measured by continuous glucose monitoring (CGM) using the Dexcom G7 sensor and point-of-care (POC) testing with the Accu-Chek device is assessed when the CGM sensor is placed in the abdomen compared to the upper arm

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Zorggroep Twente Almelo, Almelo, Overijssel
  - Deventer Ziekenhuis, Deventer, Overijssel
  - Medisch Spectrum Twente, Enschede, Overijssel

IPD SHARING:
Plan to Share IPD: No
We are committed to sharing individual participant data (IPD) in accordance with established data-sharing principles. However, access to our IPD will only be granted upon formal request. Researchers interested in obtaining the data must submit a detailed request to the study's designated contact person. This request should include a thorough explanation of the intended use of the data, the research plan, and ethical considerations. Each request will be carefully evaluated based on the proposed study's merits and alignment with our data-sharing policies before a decision is made regarding data access.